CLINICAL TRIAL: NCT01083017
Title: Interventional Prospective Cohort Study, Multi-center With Nested Case-control Studies (Family-based and Non-family Based) on Individuals With Resistant Arterial Hypertension.
Brief Title: Resistant Arterial Hypertension Cohort Study
Acronym: RAHyCo
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Georg EHRET, intern, University Hospital, Geneva
Other Study IDs: RAHyCOstudy; 33CM30-124087 (Other Grant/Funding Number: Swiss National Science Foundation); CER09-237 (Other: IRB)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Hypertension; Essential Hypertension; Resistant Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Chlorthalidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, DNA, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- chlorthalidone
  Interventions: Drug: chlorthalidone
- motivational invervention: motivational interview(s) vs. repeated calls vs. no particular intervention
  Interventions: Behavioral: motivational intervention for non-compliant individuals
- standardized anti-hypertensive treatment
  Interventions: Drug: standardized anti-hypertensive treatment

INTERVENTIONS:
Drug: chlorthalidone — chlorthalidone 25mg/d vs. chlorthalidone 50mg/d
  Groups: chlorthalidone
Behavioral: motivational intervention for non-compliant individuals — motivational interview(s) vs. repeated calls vs. no particular intervention
  Groups: motivational invervention
Drug: standardized anti-hypertensive treatment — olmesartan, amlodipine, chlorthalidone, +- spironolactone
  Groups: standardized anti-hypertensive treatment

SUMMARY:
The purpose of this study is to investigate the epidemiology of resistant hypertension, evaluate the efficacy and feasibility of a standardized drug treatment regimen (including the randomization of two doses of the diuretic used - chlorthalidone), study two interventions in the group of patients that is non-compliant, and study environmental and genetic variables of individuals with resistant hypertension in a family design.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* resistant hypertension at the moment of inclusion
* 18 years or more, both sexes are included
* women at reproductive age: consenting to use oral contraception

Exclusion Criteria:

* patients mentally impaired or unable to give informed consent
* patients speaking only a foreign language other than French, German, or English
* patients living far away, making the study visits not practical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients addressed to a speciality consultation at Geneva University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2011-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
blood pressure control | at 12 weeks after initiation of standard treatment

SECONDARY OUTCOMES:
cardiovascular morbidity and mortality | 5 years
  additional secondary: BP control at yearly follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette PECHERE, MD, Principal Investigator — Geneva University Hospitals, Switzerland; Georg B EHRET, MD, Principal Investigator — Geneva University Hospitals, Switzerland
Locations (3):
- Switzerland (3):
  - Geneva University Hospitals, Geneva
  - Lausanne University Hospital, CHUV, Lausanne
  - Kantonsspital Luzern, Lucerne